CLINICAL TRIAL: NCT04995575
Title: Dissecting the Pathways of Therapy Resistance in Early Breast Cancer: A Sub-study of the EORTC 10041/BIG 3-04 MINDACT Study
Brief Title: Dissecting the Pathways of Therapy Resistance in Early Breast Cancer
Acronym: MINDACTRelapse
Status: Terminated | Type: Observational
Why Stopped: Closed as not feasible
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-1550-BCG
Record Dates: First submitted 2019-08-07; First posted 2021-08-09 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; MINDACT; relapses; metastasis; molecular analysis; sequencing
MeSH Terms: conditions — Breast Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — tumor tissue, whole blood, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- all MINDACT patients who relapse
  Interventions: Procedure: collection of the biopsy, blood samples

INTERVENTIONS:
Procedure: collection of the biopsy, blood samples — for the patients recruited retrospectively collection of biopsy is not considered intervention, as the relapse samples were collected according to standard of care in the participating hospitals.
  For the prospective collection of samples, the relapsed patients will be asked to donate tissue and blood samples

SUMMARY:
Within the 1st step MINDACT patients who have already relapsed will be asked to participate. For these patients a biopsy of the metastasis should have been taken. A molecular analysis of the stored primary tumor sample and of the metastatic sample, using new technologies, will be performed, and the characteristics of both samples will be compared.

Within the 2nd step a prospective collection of the metastasis samples will be implemented and analysis of biological material from relapsing MINDACT patients is foreseen.

This process will provide insights on the biology of breast cancer and allow us to better understand mechanisms of resistance to therapies, contributing to overcoming this important problem.

ELIGIBILITY:
Retrospective part (part I):

* Written informed consent of agreement for participating in the research project.
* Patients must have been enrolled in the MINDACT study and received randomized or non-randomized treatment within the study, of any type and any duration and have consented for future research or are willing to provide consent for use of the primary tumour sample.
* Patients must have a local, regional or distant breast cancer relapse or new primary breast cancer lesion and have undergone a bioptic/excision procedure of the new, not previously irradiated, lesion as part of routine clinical practice before initiation of a subsequent line of systemic treatment (any line).
* At least one Formalin-Fixed Paraffin-embedded (FFPE) tissue block or fresh frozen tissue (FFT) from the biopsy or from the resection specimen of the relapsed or new primary disease site, available for translational research purposes.
* If blood or normal tissue (e.g. non tumoral) is available in the hospital, it will be collected as well. For clarity, if normal tissue is not available, patients remain eligible for the research project but will not be prioritized for the molecular analysis.
* Biopsies of bone lesions are accepted if no other metastatic lesions are available.
* Patients with brain metastases are accepted if brain-tissue is provided through surgical excision as part of the routine clinical practice.

Prospective part (part II):

* Written informed consent of agreement for participating in the research project.
* Patients must have been enrolled in the MINDACT study and received randomized or non-randomized treatment within the study, of any type and any duration and have consented for future research or are willing to provide consent for use of the primary tumour sample.
* Patients must have a new diagnosis of local, regional or distant breast cancer relapse or new primary breast cancer lesion based on physical, radiological and/or laboratory evaluation and will undergo a biopsy of this new, not previously irradiated, lesion as part of routine clinical practice.
* The biopsy of the local, regional or distant breast cancer relapse or new primary breast cancer lesion must be conducted either at the initial diagnosis of the breast cancer (BC) relapse or at the first disease progression upon any line of systemic treatment received. Of note, the biopsy of the metastatic lesion must be conducted before initiation of a subsequent line of systemic treatment.
* At least one FFPE tissue block or FFT from the biopsy or from the resection specimen of the relapsed or new primary disease site, available for translational research purposes.
* Biopsies of bone lesions are accepted if no other metastatic lesions are available.
* Patients with brain metastases are accepted if brain-tissue is provided through surgical excision as part of the routine clinical practice.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
* The patient agrees to provide blood samples at enrolment in research project and at the time of new disease progression.
* The patient is eligible if she has not received palliative radiotherapy prior to the biopsy.
* Patients who participated in the retrospective part are allowed to participate in the prospective part as long as there is another new breast cancer lesion (local, regional or distant relapse or new primary breast tumour) identified which has not been irradiated previously that will be biopsied by the site. The biopsy and blood draw should be performed prior to the start of next line of treatment.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: please see eligibility criteria as this is a 1 cohort study
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Number of enrolled patients per year with adequate clinicopathologically annotated biological material and clinical data. | 2 years after FPI
  Collection of tissue from the first site of relapse or new primary breast cancer, and blood samples for patients still alive that have relapsed (retrospective collection) or will relapse (prospective collection)
Disease progression | 2 years after FPI
  Characterization of disease progression using molecular characterization of tumour and germline molecular markers in tissue and blood.
Treatment resistance | 2 years after FPI
  Treatment resistance studies aiming to verify if a given mechanism is responsible for the relapse after exposure to anticancer agents will be performed using molecular characterization of tumour and germline molecular markers in tissue and blood..

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (4):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Institut Jules Bordet-Hopital Universitaire ULB, Brussels
  - Hopital De Jolimont, Haine-Saint-Paul
  - CHU-UCL Namur - CHU Site Sainte-Elisabeth-UCL Namur, Namur
- Ziekenhuisgroep Twente - Twenteborg Ziekenhuis (3), Almelo, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The access to the data collected within this study, upon study completion could be requested by filling in the request form on EORTC website.